CLINICAL TRIAL: NCT06278896
Title: Early Neutropenic Fever De-escalation (END) of Antibiotics Study
Brief Title: Early Neutropenic Fever De-escalation of Antibiotics Study
Acronym: END
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Lindsey R. Baden, MD, Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-684-END
Record Dates: First submitted 2024-01-03; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Hematologic Malignancy; Febrile Neutropenia; Antibiotic Stewardship
Keywords: Febrile Neutropenia
MeSH Terms: conditions — Hematologic Neoplasms; Febrile Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants will stop empiric antibiotic therapy after their episode of fever if afebrile for 48 hours, no clinically documented source of bacterial infection, and no hemodynamic or respiratory decompensation.
  Interventions: Drug: Cessation of antibiotics
- Control Arm (No Intervention): Participants will continue antibiotic therapy until count recovery and/or standard of care as deemed by inpatient providers, which is the current guidelines recommended by the IDSA.

INTERVENTIONS:
Drug: Cessation of antibiotics — Stop antibiotic therapy after episode of fever if afebrile for 48 hours, no clinically documented source of bacterial infection, and no hemodynamic or respiratory decompensation.
  Other Names: Stop antibiotics
  Arms: Intervention Arm

SUMMARY:
This is a randomized, open label clinical trial among individuals with hematologic conditions. The trial aims to evaluate the safety and clinical outcomes of de-escalating antibiotic therapy among stable individuals diagnosed with neutropenic fever, in which no bacterial infection has been identified.

DETAILED DESCRIPTION:
Background:

The Infectious Disease Society of America (IDSA) guidelines for febrile neutropenia conflict with several other international guidelines on duration of antibiotic therapy in patients with febrile neutropenia without a documented infectious source. The IDSA recommends continuing antibiotic therapy until clear signs of marrow recovery, while other guidelines, including the European guidelines, allow for earlier discontinuation if no source of bacterial infection is identified. Benefits of earlier discontinuation of antibiotics include mitigating the risk of induction and amplification of antibiotic resistance, decreased disruption of the microbiome, as well as minimizing potential side effects and complications associated with long-term antibiotic use. To date the only randomized clinical trial in adults evaluating an abridged course of antibiotic therapy in high-risk patients with febrile neutropenia (defined as neutropenia for at least 7 days) was a superiority study that demonstrated fewer days of antibiotic use in the control arm. Safety data were a secondary outcome. Further research is needed to assess the safety and clinical outcomes of targeted antibiotic therapy for patients with febrile neutropenia.

Study Design:

This is a randomized, open label clinical trial among individuals with hematologic conditions. The trial aims to evaluate the safety and clinical outcomes of de-escalating antibiotic therapy among stable individuals diagnosed with neutropenic fever, in which no bacterial infection has been identified.

Treatment Regimen:

Intervention Arm (Arm A): Stop antibiotic therapy after episode of fever if afebrile for 48 hours, no clinically documented source of bacterial infection, and no hemodynamic or respiratory decompensation.

Control Arm (Arm B): Continue antibiotic therapy per IDSA guidelines until count recovery and/or standard of care as deemed by inpatient providers.

Study Participants:

The study population will comprise adults who have hematologic high-risk neutropenia (likely > 7 days).

ELIGIBILITY:
Inclusion Criteria:

1. Participant or healthcare proxy with the ability to understand and willingness to sign an informed consent.
2. Adults >18 years old.
3. Likely to have neutropenia > 7 days including such conditions as: acute leukemia; lymphoproliferative disease; multiple myeloma; myelodysplastic syndrome; bone marrow aplasia and autologous or allogeneic hematopoietic stem cell transplantation. Neutropenia defined as absolute neutrophil count <500.
4. Received or planned to receive cytotoxic chemotherapy. No restrictions on prior therapy regarding dose or agent.
5. High-risk neutropenia defined as expected duration of absolute neutrophil count less than 500 cells/µL for seven or more days.
6. Admitted as an inpatient at Mass General Brigham or Dana Farber Cancer Institute (DFCI).
7. Initial fever (defined as a single oral temperature of ≥38.3°C or a temperature of ≥38.0°C sustained over a one-hour period) during hospital admission or as reason for admission.
8. Has been afebrile for 48 hours.

Exclusion Criteria:

1. Microbiologically or clinically suspected bacterial infection after index fever.
2. Exposure to treatment antibacterial therapy 72 hours before first fever occurrence other than antibiotics deemed as prophylaxis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Mortality, transfer to the ICU, septic shock, culture-confirmed bacteremia | 60 days
  To compare number of patients with a 60-day composite of mortality, transfer to the ICU, septic shock, culture-confirmed bacteremia in each arm.
Antibiotic utilization | 60 days
  To compare the days of antibiotic spectrum coverage (DASC), in each arm between randomization and count recovery.

SECONDARY OUTCOMES:
Mortality post F&N | 60 days
  To compare the rates of mortality within 60 days after first neutropenic fever in each arm.
Drug resistance | 60 days
  To compare the rates of acquisition of multidrug resistant gram-negative bacilli (resistant to 3 or more antibiotic classes) and vancomycin resistant enterococci within 60 days after first neutropenic fever in each arm.
Clostridium difficile infection | 60 days
  To compare the rates of Clostridium difficile infection (CDI) within 60 days after first neutropenic fever infection in each arm.
Candidiasis | 60 days
  To compare the rates of candidemia and invasive candidiasis within 60 days after first neutropenic fever in each arm.
Adverse Events | 60 days
  To compare the rates of grade 3, 4, and 5 adverse events in each arm within 60 days after first neutropenic fever.
Allergic Reactions | 60 days
  To compare the rates of allergic reactions or side effects attributed to antibiotics that required antibiotic cessation or change within 60 days after first neutropenic fever.
Bacteremia | 60 days
  To compare the rates of bacteremia within 60 days after randomization.
Neutropenia | 60 days
  To compare the rates of neutropenia at antibiotic stop date.
Length of stay | 60 days
  To compare the length of hospital stay in each arm.
Readmissions | 60 days
  To compare the rates of non-elective hospital readmission within 60 days in each arm.
Fever | 60 days
  To compare the rates of new fever after index fever in each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey R Baden, MD, Principal Investigator — Brigham and Women's Hospital, Dana Farber Cancer Institute, Harvard

IPD SHARING:
Plan to Share IPD: No